CLINICAL TRIAL: NCT04552041
Title: Multicenter Double-blind Placebo-controlled Randomized Parallel-group Clinical Trial of Efficacy and Safety of Prospekta in the Treatment of Cognitive, Behavioral and Psychiatric Disorders in Patients With Vascular Dementia.
Brief Title: Prospekta in the Treatment of Cognitive, Behavioral and Psychiatric Disorders in Patients With Vascular Dementia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-MAP-003
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-01

CONDITIONS: Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospekta (Experimental): Two tablets per intake 2 times a day (approximately at the same time), outside of meal (between meals or 15 minutes prior to meal or drinking). The tablets should be held in mouth until completely dissolved. The overall duration of treatment is 24 weeks.
  Interventions: Drug: Prospekta
- Placebo (Placebo Comparator): Two tablets per intake 2 times a day (approximately at the same time), outside of meal (between meals or 15 minutes prior to meal or drinking). The tablets should be held in mouth until completely dissolved. The overall duration of treatment is 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prospekta — Oral administration.
  Other Names: MMH-MAP
  Arms: Prospekta
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
Study purpose:

- evaluate clinical efficacy ands afety of Prospekta in the treatment of cognitive, behavioral and psychiatric disorders in patients with vascular dementia.

Study objectives:

* evaluate and compare changes in cognitive functions, in behavioral and in psychiatric dementia symptoms in Prospekta and Placebo groups after 24-weeks of treatment
* evaluate and compare the frequency, severity and causal relationship of adverse events (AEs) with the type of therapy in Prospekta and Placebo groups (including central nervous system AEs during therapy, their relationship with the study drug and other characteristics).

DETAILED DESCRIPTION:
Design: double-blind placebo-controlled randomized parallel-group clinical trial. The study will enroll male and female patients aged 60-85 years inclusively diagnosed with vascular dementia verified at Visit 1 according to the criteria of The National Institute of Neurological Disorders and Stroke National Institute of Neurological Disorders and Stroke-Association Internationale pour la Recherche et l'Enseignement en Neurosciences - NINDS-AIREN. Severity of vascular dementia should be moderate or mild (10-24 points according to Mini-Mental State Examination - MMSE), without signs of depression (total Cornell Scale for Depression in Dementia (CSDD) score ≤10).

After signing patient information sheet (informed consent form) to participate in the study, at Visit 1 (from day -14 to day 1) complaints and medical history will be collected, objective examination, recording vital signs (BP, RR, HR) will be performed and compliance of the subject's diagnosis with NINDS-AIREN vascular dementia criteria will be evaluated. The study investigator will assess cognitive disorders using Mini-Mental State Examination (MMSE) and Montreal Сognitive Assessment (МоСА). The investigator and the patient's caregiver will fill Neuropsychiatric Inventory Сlinician (NPI-С), and СSDD scales. The patient will undergo brain MRI (in the absence of brain MRI data within the previous 12 months before inclusion in the study).

Concomitant therapy and concomitant diseases and conditions will be recorded. If inclusion/exclusion criteria are met, the patient will be randomized to one of the two groups: group 1 will receive Prospekta 2 tablets twice daily; group 2 will receive Placebo using the study drug dosing regimen.

Treatment duration will be 24 weeks during which 6 Visits will be made. At visits 2 and 3 (week 4±3 days and week 8±3 days) the study investigator will make a phone call and collect the complaints, monitor the prescribed and concomitant therapy, evaluate therapeutic safety.

At visit 4 (week 12±7 days) the study investigator will collect complaints, record objective examination findings and vital signs, monitor the prescribed and concomitant therapy, evaluate therapeutic safety and compliance, dispense the study drug until the next visit. The study investigator and caregiver will fill NPI-C.

At visits 5 and 6 (week 16±3 days and week 20±3 days) the study investigator will make a phone call and collect the complaints, monitor the prescribed and concomitant therapy, evaluate therapeutic safety.

At visit 7 (week 24±7 days) the study investigator will collect complaints, perform objective examination, record vital signs, monitor the prescribed and concomitant therapy, evaluate therapeutic safety, evaluate compliance. The study investigator will fill MоСА and Clinical Global Impression Efficacy Index (CGI-EI). The study investigator and caregiver will fill NPI-C.

During the study the treatment for concomitant diseases will be allowed with the exception of the drugs specified in the section "Prohibited concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 60-85 years old inclusively.
2. Subjects with verified diagnosis of vascular dementia.
3. Presence of all the vascular dementia criteria according to NINDS-AIREN:

   A. Presence of dementia, which is defined as a decline in cognitive function relative to the previous level of functioning, manifested by impairments in memory and two or more cognitive domains (orientation, attention, language, visuospatial functions, executive functions, motor control and praxis), preferably established during a clinical trial and confirmed by neuropsychological testing.

   The cognitive impairment must be so severe that it affects daily activity, reducing it independently of the physical consequences of the stroke.

   B. The presence of cerebrovascular disease, confirmed by signs of focal damage on neurological examination, such as hemiparesis, lower facial weakness, Babinski sign, sensory deficit, hemianopsia or dysarthria associated with stroke (either a history of stroke or absence of such anamnestic information), and neuroimaging (CT or MRI) signs of cerebrovascular disease, including multiple infarcts in the territory of large vessels, or a single infarction in a strategically important area (angular gyrus, thalamus, basal ganglia, or the territory of the anterior or posterior cerebral arteries), as well as multiple lacunae in the region of the basal ganglia or white matter, or significant damage to the periventricular white matter, or a combination of the above lesions.

   C. There is an association between dementia and cerebrovascular disease as follows:
   1. onset of dementia within 3 months of stroke;
   2. sharp deterioration of cognitive functions; or fluctuating, stepwise progression of cognitive impairment.
4. Availability of permanent caregiver throughout the study (nurse or relatives).
5. Total Mini-Mental State Examination (MMSE) score - 10-24.
6. Total MoCA score <26.
7. Total NPI-C aggression and agitation domain score ≥14.
8. Аbsence of depression (total Cornell Scale for Depression in Dementia (CSDD) score ≤10).
9. Brain MRI confirming the diagnosis of vascular dementia within 1 year prior to enrollment (or brain MRI performed at enrollment visit).
10. Patients giving their consent to use reliable contraception throughout the study (for males).
11. Availability of signed patient information sheet and informed consent form for participation in the clinical trial.

Exclusion Criteria:

1. Signs of intracerebral hemorrhage, brain tumours causing dementia.
2. Alzheimer's disease, Parkinson disease, Lewy body dementia, multiple system atrophy, Jacob-Creutzfeld disease, Pick syndrome, corticobasal degeneration.
3. Injuries of head (S00-S09) associated with impaired consciousness, cerebral contusion or open craniocerebral traumas.
4. Toxicity-related dementia (including drug-induced), multiorgan failure or metabolic and toxic disorders (chronic hypothyroidism, decompensated diabetes mellitus, avitaminoses, etc.).
5. Other psychiatric diseases besides dementia: mental disorders and behavioral disorders due to use of psychoactive substances (F10-19) schizophrenia, schizotypal and delusional disorders (F20-29).
6. Mental retardation (F70-79).
7. Inflammatory lesions of the brain with persistent neurological deficit.
8. Malignant neoplasms.
9. Previously diagnosed cardiovascular diseases with functional class IV (according to New York Heart Association, 1964).
10. Unstable angina pectoris, myocardial infarction or ischemic stroke within the last 6 months.
11. Female patients with childbearing potency.
12. Allergy/intolerance of any of the study drugs components including secondary to lactase deficiency.
13. Any conditions which, according to the investigator opinion, may interfere with the patient's participation in the study.
14. History of treatment noncompliance, mental diseases, alcoholism or drug abuse which will prevent from following the study procedures, according to investigator's opinion.
15. Participation in clinical trials for 3 months prior to enrollment in this study.
16. Use of any medications specified in "Prohibited concomitant medications" within 1 month before enrollment.
17. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
18. Patients who work for OOO "NPF "Materia Medica Holding" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kamchatnov, professor, Principal Investigator — V.M. Buyanov Moscow City Clinical Hospital, Moscow, Russia
Locations (33):
- Russia (33):
  - Northern State Medical University/Department of Family Medicine and Internal Medicine, Arkhangelsk
  - Belgorod Regional Clinical Hospital of St. Joasaph/Neurological department, Belgorod
  - Hospital "Russian Railways - Medicine" of the city of Bryansk/Medical rehabilitation department, Bryansk
  - Engels Psychiatric Hospital, Engel's
  - Kazan State Medical University/Department of Neurology and Rehabilitation, Kazan'
  - City Clinical Hospital named after V.M. Buyanov of the Moscow City Health Department/1st neurological department, Moscow
  - Peoples' Friendship University of Russia/Department of Psychiatry, Psychotherapy and Psychosomatic Pathology, Moscow
  - Central Clinical Hospital of the Russian Academy of Sciences/Treatment and Diagnostic Center, Moscow
  - Psychiatric hospital # 1 named after P.P. Kashchenko, Nikol’skoye
  - Privolzhsky Research Medical University/Department of Medical Rehabilitation, Nizhny Novgorod
  - Nizhny Novgorod Regional Clinical Hospital. N. A. Semashko/Outpatient department, Nizhny Novgorod
  - Orenburg Regional Clinical Psychiatric Hospital # 1/Psychoneurological dispensary, Orenburg
  - Pyatigorsk City Clinical Hospital # 2/Neurological department, Pyatigorsk
  - LLC "Treatment and reabilitation research center " PHOENIX "/Day hospital # 1, Rostov-on-Don
  - Psychoneurological dispensary # 10/Medical rehabilitation department, Saint Petersburg
  - St. Nicholas Psychiatric Hospital, Saint Petersburg
  - St. Petersburg Research Institute of Emergency Medicine named after I.I. Janelidze/Medical Rehabilitation Department, Saint Petersburg
  - Leningrad Regional Clinical Hospital/Neurological department, Saint Petersburg
  - Psychoneurological dispensary # 5/Day hospital, Saint Petersburg
  - Samara City Clinical Hospital # 1 named after N.I. Pirogov/Neurological department for patients with cerebrovascular accident # 24, Samara
  - Saratov State Medical University V. I. Razumovsky/Department of Neurology named after K.N. Tretyakov, Saratov
  - City Clinical Hospital # 2 named after V.I. Razumovsky, Saratov
  - Saratov City Psychoneurological Dispensary, Saratov
  - Regional Clinical Psychiatric Hospital of St. Sophia, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - Stavropol Regional Clinical Specialized Psychiatric Hospital # 1/Somatogeriatric department #19, Stavropol
  - Republican Clinical Hospital named after G.G. Kuvatov, Ufa
  - Bashkir State Medical University/Department of Neurology, Ufa
  - Ulyanovsk Regional Clinical Hospital/Outpatient department, Ulyanovsk
  - Regional Clinic Hospital, Vladimir
  - Volgograd State Medical University/Department of Neurology, Neurosurgery with the Course of Medical Genetics, Volgograd
  - Vsevolozhsk clinical interdistrict hospital/Neurological department, Vsevolozhsk
  - Sverdlovsk Regional Clinical Psychiatric Hospital, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 406 patients signed informed consent, of which 7 patients did not pass the screening.
Groups:
- Prospekta: Two tablets per intake 2 times a day (approximately at the same time), outside of meal (between meals or 15 minutes prior to meal or drinking). The tablets should be held in mouth until completely dissolved.
  Prospekta: Oral administration.
- Placebo: Two tablets per intake 2 times a day (approximately at the same time), outside of meal (between meals or 15 minutes prior to meal or drinking). The tablets should be held in mouth until completely dissolved.
  Placebo: Oral administration.
Period: Overall Study
Arm/Group | Prospekta | Placebo
Started | 204 | 195
Completed | 204 | 195
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospekta | Placebo | Total
Number analyzed (Participants) | 204 | 195 | 399
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 173 | 163 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.0) | 72.7 (6.9) | 72.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 141 | 290
  Male | 55 | 54 | 109
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 204 | 195 | 399

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Montreal Сognitive Assessment (MoCA) Score
Description: MoCA is the test for assessment of cognitive impairment. The score ranges between 0 and 30. A score of 26-30 is normal. A score less than 26 is considered as mild cognitive impairment. Higher values represent a better outcome.
Time Frame: Baseline, 24 weeks
Population: 10 patients from Prospekta group and 7 patients from Placebo group were excluded from the trial before 24 week therefore no data was collected on 24 weeks timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 204 | 195
score on a scale
  Baseline | 17.0 (3.6) | 17.3 (3.7)
  After 24 weeks: number analyzed (Participants) | 194 | 188
  After 24 weeks | 20.5 (4.7) | 19.2 (4.9)
  ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 188
  ∆ between baseline and 24 weeks | 3.3 (3.1) | 1.9 (3.1)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 24 weeks row; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Mean Neuropsychiatric Inventory-Clinician (NPI-С) Score
Description: NPI-C allows to evaluate severity of behavioural and mental disorders associated with dementia. The scale consists of 14 domains. Scoring for "delusional ideas" (8 items) is 0-24 points, for "hallucinations" (7 items) - 0-21, "agitation" (13 items) - 0-39, "aggression" (8 items) - 0-24, "dysphoria" (13 items) - 0-39, "anxiety" (14 items) - 0-42, "euphoria" (6 items) - 0-18, "apathy" (11 items) - 0-33, "disinhibition" (16 items) - 0-48, "irritability" (12 items) - 0-36 , "aberrant motor behaviour" (9 items) - 0-27, "sleep disorders" (8 items) - 0-24, "appetite disorders" (9 items) - 0-27, "aberrant vocalizations" (8 items) - 0-24. Each item is rated for frequency (a 4-point scale from 1 [occasionally] to 4 [very frequent]) and severity (a 3-point scale from 1 [mild] to 3 [marked]). The total NPI score is the frequency ratings multiplied by the severity ratings. Total maximum score for all domains is 426 (higher score indicates worse outcome).
Time Frame: Baseline, 24 weeks
Population: 8 patients from Prospekta group and 6 patients from Placebo group were excluded from the trial before 24 week therefore no data was collected on 24 weeks timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 204 | 195
score on a scale
  Baseline: number analyzed (Participants) | 202 | 195
  Baseline | 57.0 (26.7) | 55.5 (25.5)
  After 24 weeks: number analyzed (Participants) | 194 | 189
  After 24 weeks | 39.8 (23.6) | 42.8 (27.6)
  ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  ∆ between baseline and 24 weeks | -17.1 (15.1) | -13.0 (15.1)
  Domain "Delusional ideas" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Delusional ideas" ∆ between baseline and 24 weeks | -0.2 (0.9) | -0.1 (0.6)
  Domain "Hallucinations" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Hallucinations" ∆ between baseline and 24 weeks | -0.1 (0.4) | -0.0 (0.5)
  Domain "Agitation" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Agitation" ∆ between baseline and 24 weeks | -4.2 (3.9) | -3.6 (4.3)
  Domain "Aggression" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Aggression" ∆ between baseline and 24 weeks | -2.0 (2.3) | -1.8 (2.3)
  Domain "Dysphoria" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Dysphoria" ∆ between baseline and 24 weeks | -1.7 (3.1) | -1.3 (3.5)
  Domain "Anxiety" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Anxiety" ∆ between baseline and 24 weeks | -2.3 (3.8) | -1.6 (3.4)
  Domain "Euphoria" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Euphoria" ∆ between baseline and 24 weeks | -0.1 (0.7) | -0.2 (1.0)
  Domain "Apathy" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Apathy" ∆ between baseline and 24 weeks | -1.1 (3.6) | -0.6 (4.0)
  Domain "Disinhibition" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Disinhibition" ∆ between baseline and 24 weeks | -0.5 (2.1) | -0.4 (1.6)
  Domain "Irritability" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Irritability" ∆ between baseline and 24 weeks | -2.1 (3.9) | -1.7 (3.2)
  Domain "Aberrant motor behaviour" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Aberrant motor behaviour" ∆ between baseline and 24 weeks | -0.6 (1.4) | -0.1 (1.2)
  Domain "Sleep disorders" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Sleep disorders" ∆ between baseline and 24 weeks | -1.5 (2.4) | -1.2 (2.4)
  Domain "Appetite disorders" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Appetite disorders" ∆ between baseline and 24 weeks | -0.3 (1.4) | -0.1 (1.1)
  Domain "Aberrant vocalizations" ∆ between baseline and 24 weeks: number analyzed (Participants) | 194 | 189
  Domain "Aberrant vocalizations" ∆ between baseline and 24 weeks | -0.3 (0.9) | -0.2 (1.0)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0028, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Prospekta vs Placebo; This analysis applies to domain "Delusional ideas" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.1739, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Prospekta vs Placebo; This analysis applies to domain "Hallucinations" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0559, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Prospekta vs Placebo; This analysis applies to domain "Agitation" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0174, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Prospekta vs Placebo; This analysis applies to domain "Aggression" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.3330, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Prospekta vs Placebo; This analysis applies to domain "Dysphoria" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.1037, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Prospekta vs Placebo; This analysis applies to domain "Anxiety" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0329, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Prospekta vs Placebo; This analysis applies to domain "Euphoria" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.2700, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Prospekta vs Placebo; This analysis applies to domain "Apathy" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0557, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Prospekta vs Placebo; This analysis applies to domain "Disinhibition" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.9820, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Prospekta vs Placebo; This analysis applies to domain "Irritability" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.4626, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Prospekta vs Placebo; This analysis applies to domain "Aberrant motor behaviour" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0006, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Prospekta vs Placebo; This analysis applies to domain "Sleep disorders" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.3725, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Prospekta vs Placebo; This analysis applies to domain "Appetite disorders" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.1013, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Prospekta vs Placebo; This analysis applies to domain "Aberrant vocalizations" ∆ between baseline and 24 weeks row; Test type: Superiority; p = 0.0432, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Mean Montreal Сognitive Assessment (MoCA) Score
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: 8 patients from Prospekta group and 7 patients from Placebo group were excluded from the trial before 12 week therefore no data was collected on 12 weeks timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 204 | 195
score on a scale
  Baseline | 17.0 (3.6) | 17.3 (3.7)
  After 12 weeks: number analyzed (Participants) | 196 | 188
  After 12 weeks | 19.1 (4.1) | 18.9 (4.2)
  ∆ between baseline and 12 weeks: number analyzed (Participants) | 196 | 188
  ∆ between baseline and 12 weeks | 2.0 (2.2) | 1.6 (2.2)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 12 weeks row; Test type: Superiority; p = 0.0316, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Mean Neuropsychiatric Inventory-Clinician (NPI-С) Score
Description: as for outcome 2
Time Frame: Baseline, 12 weeks
Population: 7 patients from Prospekta group and 7 patients from Placebo group were excluded from the trial before 12 week therefore no data was collected on 12 weeks timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 204 | 195
score on a scale
  Baseline: number analyzed (Participants) | 202 | 195
  Baseline | 57.0 (26.7) | 55.5 (25.5)
  After 12 weeks: number analyzed (Participants) | 196 | 188
  After 12 weeks | 47.0 (24.3) | 47.1 (24.4)
  ∆ between baseline and 12 weeks: number analyzed (Participants) | 195 | 195
  ∆ between baseline and 12 weeks | -10.5 (15.5) | -8.1 (11.8)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to ∆ between baseline and 12 weeks row; Test type: Superiority; p = 0.1483, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mean Clinical Global Impression Efficacy Index (СGI-EI) Score
Description: Indicators of therapeutic and side effects, efficacy index on the scale of the general clinical impression CGI-EI (Clinical Global Impression Scale - Efficacy Index) after 24 weeks from the start of study therapy. Evaluation of the response to treatment should take into account both therapeutic efficacy and treatment-related side effects. Side effects value from 1 to 4. Therapeutic effect value as 0,4,8 or 12 points. The efficacy index is a sum. The minimum value is 1, the maximum value is 16. A lower score on the scales is the best outcome.
Time Frame: After 24 weeks of the treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prospekta | Placebo
Number analyzed (Participants) | 204 | 195
score on a scale
  Therapeutic effect | 2.4 (0.9) | 2.1 (0.8)
  Side effects | 1.1 (0.3) | 1.1 (0.2)
  Efficiency Index | 2.3 (0.9) | 2.0 (0.8)
Statistical Analysis 1: Comparison: Prospekta vs Placebo; This analysis applies to Therapeutic effect row; Test type: Superiority; p = 0.0018, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Prospekta vs Placebo; This analysis applies to Side effects row; Test type: Superiority; p = 0.4733, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Prospekta vs Placebo; This analysis applies to Efficiency index row; Test type: Superiority; p = 0.0035, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Registration of AEs begins after taking the first dose of the study drug, continues throughout the entire period of study therapy - 24 weeks, as well as for 24 hours after the last dose of the study drug.
Arm/Group | Prospekta | Placebo
All-Cause Mortality (participants affected / at risk) | 2/204 | 0/195
Serious Adverse Events (participants affected / at risk) | 6/204 | 2/195
Other Adverse Events (participants affected / at risk) | 61/204 | 52/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospekta (N=204) | Placebo (N=195)
Pneumonia caused by coronavirus infection COVID-19 (Infections and infestations) | 4 (4) | 2 (2)
Progressive angina (Cardiac disorders) | 1 (1) | 0 (0)
Cardioembolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospekta (N=204) | Placebo (N=195)
Pancreatic tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis, worsening (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive hemorrhagic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral respiratory tract infection (Infections and infestations) | 7 (7) | 4 (4)
Coronavirus infection COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Laboratory confirmed coronavirus infection COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Exacerbation of chronic bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Exacerbation of cystitis (Infections and infestations) | 1 (1) | 0 (0)
Acute upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Acute rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia caused by coronavirus infection COVID-19 (Infections and infestations) | 4 (4) | 2 (2)
Cold (Infections and infestations) | 1 (1) | 0 (0)
Chronic rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Increased blood pressure (Investigations) | 6 (6) | 7 (7)
Increased body temperature (Investigations) | 1 (1) | 0 (0)
Lower blood pressure (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decompensated diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired fasting glycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Bronchitis, chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bleeding from the paranasal sinus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension functional class II according to WHO classification (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post-vaccination reaction (Immune system disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria-like rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypochromic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chronic iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain, exacerbation (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Ankle hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Degenerative spinal disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness of the lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis, exacerbation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness of the lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carotid atheroma (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 16 (16)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tension type headache (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9) | 12 (12)
Dyscirculatory encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Daytime sleepiness (Nervous system disorders) | 1 (1) | 1 (1)
Ischialgia at the stage of exacerbation (Nervous system disorders) | 1 (1) | 0 (0)
Cardioembolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Sour taste (Nervous system disorders) | 1 (1) | 0 (0)
Cephalgia (Nervous system disorders) | 1 (1) | 0 (0)
Episodic headache (Nervous system disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease, stage 3 (Renal and urinary disorders) | 1 (1) | 0 (0)
Heart valve insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Post-infarction cardiosclerosis (Cardiac disorders) | 1 (1) | 0 (0)
Persistent atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Progressive angina (Cardiac disorders) | 1 (1) | 0 (0)
NYHA class II heart failure (Cardiac disorders) | 2 (2) | 2 (2)
Angina pectoris class II according to the Canadian classification of angina (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Arterial hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (1)
Pain at the vaccination site (General disorders) | 0 (0) | 2 (2)
Localized pain (General disorders) | 0 (0) | 1 (1)
Local edema (General disorders) | 0 (0) | 1 (1)
General weakness (General disorders) | 6 (6) | 2 (2)
Weakness (General disorders) | 4 (4) | 3 (3)
Wobbly gait (General disorders) | 0 (0) | 2 (2)
Aggressiveness (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression, exacerbation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucinatory condition (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disturbance (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Early awakening (Psychiatric disorders) | 0 (0) | 1 (1)
Lower mood (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety during medical manipulation/procedure (Psychiatric disorders) | 1 (1) | 0 (0)
Bimalleolar fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unspecified hand burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Burn of unspecified degree to unspecified area of the hand
Unspecified burn of forearm (Psychiatric disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left foot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incised wound of the left thumb (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Abrasions (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wasp sting (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bruise in the shoulder joint (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruised ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Knee contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04552041/Prot_SAP_000.pdf